CLINICAL TRIAL: NCT02439437
Title: Targeted Pain Coping Skills Training (PCST) for Prevention and Treatment of Persistent Post-Mastectomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00055890
Record Dates: First submitted 2015-03-06; First posted 2015-05-08 (Estimated); Last update posted 2020-05-01 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Psychosocial Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Psychosocial Intervention (Active Comparator): Telephone-based psychosocial intervention involving Eight telephone encounters. Each encounter will focus on strategies for dealing with pain and stress, and how to apply these strategies to patients own experiences.
  Interventions: Behavioral: Psychosocial Intervention
- Treatment as usual (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: Psychosocial Intervention — Telephone-based psychosocial intervention involving Eight telephone encounters. Each encounter will focus on strategies for dealing with pain and stress, and how to apply these strategies to patients own experiences.
  Arms: Psychosocial Intervention

SUMMARY:
This study looks at whether a coping skills training program can help women manage pain and stress after breast surgery, and lower the risk of developing chronic pain. This coping skills program includes eight training sessions that are done by telephone. These sessions will focus on strategies for dealing with pain and stress, and how to apply these strategies to subjects' own experiences.

DETAILED DESCRIPTION:
Persistent pain following breast cancer surgery is increasingly being recognized as an important clinical and public health issue due to the large numbers of women affected, the negative impact that persistent pain has on emotional and physical functioning, and its financial cost. Most of the 230,000 women that are expected to be newly diagnosed with breast cancer in the U.S. this year will undergo surgical treatment. Surgical removal of the affected breast (mastectomy) or excision of the tumor (lumpectomy) followed by radiation markedly reduces the risk of disease progression and mortality. However, women undergoing even the more limited lumpectomy are at substantial risk for persistent pain. Estimates of pain's prevalence range from 25-60% across multiple studies, with rates differing based on the stringency of the definition of persistent pain. In one recent study, 32.5% of the women who had undergone breast cancer surgery reported clinically significant persistent pain, defined as a 3/10-pain severity rating for the breast, axilla, side, or arm.

Unlike acute post-operative pain, which is considered to be a normal response to surgical trauma, persistent pain has little biological utility and has proven difficult to treat once established. A critical question is whether there are modifiable factors that contribute to the risk of developing persistent pain following breast cancer surgery that could be targeted for early, preventative intervention. To date, attempts to reduce the risk of persistent pain have focused on alterations in medical/surgical procedures; these studies have had mixed results, consistent with mixed findings in the broader literature regarding the status of medical/surgical variables as risk factors for persistent pain. In contrast, there have been multiple studies showing associations between pain catastrophizing, depression, and anxiety and persistent pain. In these studies, pain catastrophizing shows the strongest and most consistent relationship to persistent pain as evidenced in a recent meta-analysis. Consistent with the biopsychosocial theory of pain, there is also evidence from quantitative sensory testing (QST) studies that alterations in central pain modulation pathways contribute to the development of post-surgical persistent pain, including recent studies with breast cancer patients. Since pain catastrophizing has been found to be associated with pernicious alterations in central pain modulation intervening to reduce catastrophizing may be a particularly effective prevention strategy for persistent pain following breast cancer surgery. Pain coping skills training (PCST) interventions based on cognitive-behavioral principles are the only interventions demonstrated to reduce catastrophizing, alter central modulation of pain and reduce chronic pain.

The overarching hypothesis for the proposed pilot study (N=60) is that a targeted PCST protocol specifically designed for women at risk for persistent pain following breast cancer surgery (pain score of 3 or greater [0-10 scale] during the first 9 months post-surgery) will significantly reduce this devastating consequence of treatment compared to usual care with printed education materials.

Aim 1: To use a pilot RCT (N=60) to examine the feasibility, acceptability, and engagement in the targeted PCST protocol. Feasibility will be assessed by examining overall accrual, attrition, and adherence to the study protocol, engagement will be assessed by the use of intervention sessions and questionnaires (number completed), and acceptability will be assessed with a standardized measure of satisfaction.

Aim 2: To obtain an estimate of the effect size of the targeted PCST protocol for persistent post-surgical pain in comparison to the usual care condition. Effect sizes for group differences on pain burden, symptoms of anxiety and depression, breast cancer specific distress, perceived stress, sleep, interference with daily activities, pain catastrophizing, and hypothesized changes in peripheral sensitivity and central inhibition will also be computed.

The proposed study represents the next critical step in research examining persistent pain after surgical treatment for breast cancer. The proposed study will provide the necessary preliminary data for larger studies aimed at testing the targeted PCST intervention. This study will also provide preliminary data for future studies focused on pain sensitivity and central pain modulation in breast cancer survivors

ELIGIBILITY:
Inclusion Criteria:

1. prior diagnosis of Stage 0 to Stage III breast cancer
2. received first breast surgery of total or partial mastectomy within the previous 9 months
3. report average pain >/= 3 during the first 9 months after surgery on the Breast Cancer Pain Questionnaire
4. with sufficient ability to communicate in English in order to provide informed consent and complete study procedures and materials.

Exclusion Criteria:

1. < 21 years of age
2. history of prior breast cancer surgery
3. cognitive impairment documented in the medical record
4. unable to provide meaningful consent

Ages: 21 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-10-08 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Change in Pain Burden | 0 month, mid intervention(at 6 weeks), post intervention( 3 months) and 6 months
  The investigators will use BCPQ (Brest Cancer Pain Questionnaire) questionnaire to record breast pain

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca A Shelby, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States